CLINICAL TRIAL: NCT02676427
Title: Fluid Responsiveness in Septic Shock Evaluated by Caval Ultrasound Doppler Examination - "FRIEND Study"
Brief Title: Fluid Responsiveness in Septic Shock Evaluated by Caval Ultrasound Doppler Examination
Acronym: FRIEND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martin Balik, A/Prof, MD, PhD, Charles University, Czech Republic
Other Study IDs: 530/15 S-IV
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Septic Shock; Vein Collapsibility; Intravascular Doppler; Volume Responsiveness in Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: passive leg raising — passive leg raising under echocardiographic monitoring with intravascular doppler in place

SUMMARY:
The study aims at clarification of venous collapsibility measures with real venous flow measurements during dynamic maneuver testing fluid responsiveness in septic shock patients.

DETAILED DESCRIPTION:
Sedated and mechanically ventilated patients in septic shock will be enrolled in the study. A fine catheter with ultrasound doppler probe will be introduced into the central venous catheter already in place in superior vena cava. Doppler signal will be evaluated by console prototype (NILUS Medical) and continuous analysis of blood flow velocity respiratory variation will be performed. These values will be compared to standard hemodynamic monitoring parameters (central venous and arterial pressures) and to parameters acquired by transoesophageal (TOE) and transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* patients in severe sepsis or septic shock
* intubation and mechanical ventilation
* sedated patient without spontaneous respiratory efforts
* central venous catheter in place inserted via right internal jugular vein
* signed informed consent by family members

Exclusion Criteria:

* superior vena cava vascular anomaly
* irradiation of neck or mediastinum in medical history
* thrombosis of superior vena cava in medical history
* atrial fibrillation or other irregular rhythm
* permanent or external pacemaker
* aggressive mechanical ventilation (PEEP above 10 cm H2O, Pmax above 30 cm H2O)
* TOE contraindication (oesophageal varices, stricture, tumour, upper gastrointestinal bleeding)
* Pericardial effusion, constrictive pericarditis
* Moderate or severe valvular lesion
* Severe systolic dysfunction of the left (EF less than 30%) or right ventricle (FAC less than 25%)
* Intraabdominal pressure above 20 mmHg
* Open chest
* Obvious severe hypovolemia ( LVEDA<5.5cm2/m2BSA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 Years and older, mechanically ventilated ICU patients in septic shock
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | through the study, data collection during 1 year
  Evaluation of fluid responsiveness, defined as 15% increase of cardiac output after reversible fluid challenge (using PLR - passive leg raise maneuver), by ultrasound doppler evaluation of superior vena caval blood flow respiratory variation.

SECONDARY OUTCOMES:
Change of flow | through the study, data collection during 1 year
  Evaluation of fluid responsiveness by measuring a change of blood flow velocity after PLR maneuver.
Respiratory variation of flow velocity | through the study, data collection during 1 year
  Evaluation of fluid responsiveness by measuring respiratory variation of blood flow velocity in left ventricular outflow tract after PLR maneuver
Respiratory collapsibility | through the study, data collection during 1 year
  Evaluation of fluid responsiveness by measuring respiratory collapsibility of inferior vena cava after PLR maneuver.
Respiratory collapsibility | through the study, data collection during 1 year
  Evaluation of fluid responsiveness by measuring respiratory collapsibility of superior vena cava after PLR maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anaesthesia and Intensive Care, General University Hospital, 1st Medical Faculty, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No